CLINICAL TRIAL: NCT06059040
Title: Effect of Eliminating Routine Gastric Residual Volume Monitoring on Ventilator-associated Events in Patients Receiving Enteral Feeding
Brief Title: Effect of Eliminating Gastric Residual Volume Monitoring on Ventilator Associated Events
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: elimination GRV monitor on VAE
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: A parallel randomized controlled design will be used in this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention groups (Active Comparator): Patients in the intervention group will not be monitored for GRV (no GRV monitoring) and will be evaluated for the presence of feeding intolerance indicators such as vomiting, regurgitation, and abdominal distention.
  Interventions: Procedure: eliminating gastric residual volume monitoring
- control group (No Intervention): Patients in the control group will be subjected to GRV monitoring (with GRV monitoring).

INTERVENTIONS:
Procedure: eliminating gastric residual volume monitoring — eliminating gastric residual volume monitoring from routine care
  Arms: intervention groups

SUMMARY:
The aims of this study are to investigate the effect of eliminating routine GRV monitoring on VAEs in patients receiving MV and early EF, Determine the effect of eliminating routine GRV monitoring on nutritional adequacy in patients receiving MV and early EF and evaluate the effect of eliminating routine GRV monitoring on feeding intolerance in patients receiving enteral feeding.

DETAILED DESCRIPTION:
Early enteral nutrition (EN) is consistently recommended as first line nutrition therapy in critically ill patients since it favorably alters outcome, providing both nutrition and non-nutrition benefits. However, critically ill patients receiving mechanical ventilation (MV) are at risk for regurgitation, pulmonary aspiration, and eventually ventilator-associated pneumonia (VAP). EN may increase these risks when gastrointestinal (GI) dysfunction is present. Gastric residual volume (GRV) is considered a surrogate parameter of GI dysfunction during the progression of enteral feeding in the early phase of critical illness and beyond. About 62% of critically ill patients receive enteral nutrition (EN) and in patients on MV, enteral feeding was connected to a threefold increase in the development of VAP.

A new surveillance definition of ventilator-associated events (VAE) was introduced by the National Healthcare Safety Network (NHSN) in 2013 to identify patients who develop complications of MV. It outlines the various events in a step-by-step fashion, beginning with ventilator-associated complications (VAC), moving on to infectious complications (IVAC), and finally VAP. According to the NHSN, VAEs occur within 9% to 40% of mechanically ventilated patients

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged≥18 years)
* Newly admitted mechanically ventilated patients who are attached to a mechanical ventilator for at least 48 hours.
* Starting enteral nutrition via a nasogastric tube within 36 hours after intubation.

Exclusion Criteria:

* Abdominal surgery within the past month.
* History of esophageal, duodenal, pancreatic, or gastric surgery.
* Bleeding from the esophagus, stomach, or bowel.
* Enteral nutrition via a jejunostomy or gastrostomy.
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
eliminating gastric residual volume monitoring on ventilator associated events | 3 month
  use centers for disease control and prevention (CDC) calculators for evaluating VAE version 9.0 2021

SECONDARY OUTCOMES:
eliminating gastric residual volume monitoring on nutritional adequacy | 3 month
  evaluation daily caloric requirement by body mass index that calculated using the equation (Weight in kg /height in cm) 2
eliminating gastric residual volume monitoring on incidence of feeding intolerance indicators | 3 month
  evaluation of abdominal circumference, abdominal distension, bowel sounds, the episodes of vomiting and diarrhea

REFERENCES:
- [Background] Yasuda H, Kondo N, Yamamoto R, Asami S, Abe T, Tsujimoto H, Tsujimoto Y, Kataoka Y. Monitoring of gastric residual volume during enteral nutrition. Cochrane Database Syst Rev. 2021 Sep 27;9(9):CD013335. doi: 10.1002/14651858.CD013335.pub2. PMID 34596901
- [Background] Reignier J, Mercier E, Le Gouge A, Boulain T, Desachy A, Bellec F, Clavel M, Frat JP, Plantefeve G, Quenot JP, Lascarrou JB; Clinical Research in Intensive Care and Sepsis (CRICS) Group. Effect of not monitoring residual gastric volume on risk of ventilator-associated pneumonia in adults receiving mechanical ventilation and early enteral feeding: a randomized controlled trial. JAMA. 2013 Jan 16;309(3):249-56. doi: 10.1001/jama.2012.196377. PMID 23321763
- [Background] Wang Z, Ding W, Fang Q, Zhang L, Liu X, Tang Z. Effects of not monitoring gastric residual volume in intensive care patients: A meta-analysis. Int J Nurs Stud. 2019 Mar;91:86-93. doi: 10.1016/j.ijnurstu.2018.11.005. Epub 2019 Jan 3. PMID 30677592